CLINICAL TRIAL: NCT04794036
Title: Efficacy of an Asynchronous Telerehabilitation Programme in Post-COVID-19 Patients: a Feasibility Study
Brief Title: Efficacy of an Asynchronous Telerehabilitation Programme in Post-COVID-19 Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad San Jorge (Other)
Collaborators: Hospital Real Nuestra Señora de Gracia (Unknown); Hospital Royo Villanova (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: COVID-19_TRHB
Record Dates: First submitted 2021-03-01; First posted 2021-03-11 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2022-03

CONDITIONS: Coronavirus; Fatigue; Musculoskeletal Complication
Keywords: Coronavirus; Telerehabilitation; Exercise Therapy; Education
MeSH Terms: conditions — Coronavirus Infections; Fatigue

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Telerehabilitation asynchronous programme at home
  Interventions: Other: Asynchronous telerehabilitation programme
- Control Group (Active Comparator): Rehabilitation programme with an explanatory booklet at home
  Interventions: Other: Rehabilitation programme

INTERVENTIONS:
Other: Asynchronous telerehabilitation programme — Home-based physical rehabilitation programme using a telerehabilitation platform
  Arms: Experimental Group
Other: Rehabilitation programme — Home-based physical rehabilitation programme by means of an explanatory booklet
  Arms: Control Group

SUMMARY:
SARS-CoV-2 is the coronavirus responsible for developing the disease known as COVID-19. Its evolution can range from an asymptomatic course, to rapidly evolve and cause an acute respiratory syndrome. In addition to respiratory symptoms, is also has an impact on the neuromuscular systems. Therefore, the additional inactivity for hospitalization, negatively influences the loss of muscular, cardiovascular and metabolic fitness. In view of this, it is recommended that early post-acute rehabilitation be continued after the hospital phase to increase levels of physical activity, which can also be continued with long-term telerehabilitation.

This project would offer a free service of asynchronous physical telerehabilitation for the patient that is easy to implement and follow up.

For this purpose, patients will be recruited at the time of discharge from the Hospital Provincial Nuestra Señora de Gracia (HPNSG) and the Hospital Royo Villanova (HRV) in Zaragoza and two intervention groups with the same physical therapy and educational programme will be carried out. The experimental group will be carried out by means of home telerehabilitation, while the control group will receive the programme in an explanatory booklet.

The main objective is to analyse the preliminary efficacy on physical fitness of a 12-week physical therapy and therapeutic education programme using asynchronous telerehabilitation in post-COVID-19 patients, and to compare its effects with patients who have undergone the same programme, but in a non-telematic format.

The secondary objective is to analyze the feasibility of a physical home-based asynchronous telerehabilitation programme in post-COVID-19 patients.

Hypothesis: the implementation of a 12-week programme of physical therapy and therapeutic education using asynchronous telerehabilitation software is feasible and preliminarily effective in increasing physical fitness as well as adherence to treatment, and in the improvement of psychosocial factors.

DETAILED DESCRIPTION:
At the first phase, an observational study aims to investigate the physical and psychological status of patients after hospital discharge.

At the second phase, a feasibility pilot study with a single-blinded randomized clinical trial design with volunteer patients admitted to hospital and recruited at the time of discharge by COVID-19 will evaluate a physiotherapy programme. There will be an intervention group (asynchronous telerehabilitation at home) and a control group (home rehabilitation by means of an explanatory leaflet). The intervention will be carried out for 12 weeks with a follow-up at 3 and 6 months.

Intervention:

The physical rehabilitation programme will be designed with three levels of intensity of aerobic, strength and respiratory exercises, and a list of recommendations for self-management of the sequelae of the COVID-19.

The intervention will last for a total of 12 weeks at home (three days a week for 45-60 minutes a day) with a biweekly phone check-up.

All patients will be provided with the same physical rehabilitation and educational programme, with each allocation group differing in the format of the prescription.

Experimental group

A programme with exercise videos and health recommendations will be prescribed through a telerehabilitation platform to improve fatigue and fitness resulting from COVID-19. The application will be installed on patients' mobile phones and its use will be explained to them so that they can carry out the programme from their homes.

Control group The control group will receive a paper booklet with clear pictures and descriptions of the exercise and educative programme to improve fatigue and fitness.

Assessment:

Fatigue will be assessed with the fatigue severity scale (FSS). Functional capacity will be measured through operation: with the Post-COVID Functional Status Scale (PCFS), the strength with the 30" sit-to-stand (STST), the 30" arm curl test (ACT), and through aerobic capacity with de six minutes walking test (6MWT).

Psychosocial factors will be measured with the general self-efficacy scale (GSES), the depression and anxiety scale (DASS-21), the behavioral regulation questionnaire in sport (BRSQ) and the multidimensional scale of perceived social support (MSPSS).

Quality of life will be measured with the quality of life scale (SF-12).

Adherence and engagement be measured by diary recording and satisfaction with a brief interview.

Outcome measures:

Fatigue, functional status post-COVID-19, strength, aerobic capacity, anxiety and depression, behavior in sport, perceived social support and quality of life will be evaluated before intervention, after intervention (12 weeks) at 3 and 6 months for follow-up.

Adherence and satisfaction will be evaluated after intervention (12 weeks) and during intervention (each 15 days).

ELIGIBILITY:
Inclusion Criteria:

* Age range 18-75 years.
* Patients who have been hospitalized for more than 5 days for COVID-19.
* Patients who have been discharged from the hospital and present a fatigue score higher than 4 points on average on the fatigue severity scale (FSS).
* Independent walking, even with the use of any technical aid.
* Have signed the informed consent form.

Exclusion Criteria:

* Patients with central and/or peripheral neurological diseases that prevent the programme from being followed.
* Patients with rheumatic pathology or acute musculoskeletal injury in their medical history.
* Patients with severe respiratory failure: SaO2 less than 90% or respiratory rate >30.
* Patients with cardiac comorbidities or signs of cardiovascular inestability as uncontrolled arrythmia, blood pressure and/or effort angina.
* Patients with other contraindicated pathology for moderate-intensity aerobic or strength exercise.
* Patients without access to mobile internet or computer with internet at home.
* Patients with a score ≤24 on the Mini-Cognitive Examination (MEC).
* Patients who are unable to follow oral and written instructions in Spanish.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-04-05 (Actual); Primary Completion 2022-06-13 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Fatigue Severity Level | Pre-intervention (day 1); after intervention (day 84); follow up 1 (3 months after intervention); follow up 2 (6 months after intervention).
  Change in fatigue severity level. Fatigue will be assessed with the Fatigue Severity Scale (FSS). The Fatigue Severity Scale is a self-reported scale composed of 9 items. Each item is rated from 1 to 7 (from 1=strongly disagree to 7=strongly agree). In the FSS, a mean of less than 4 points is considered to be no fatigue and more than 4 is considered to present fatigue. The higher the score, the greater the severity of fatigue.

SECONDARY OUTCOMES:
Adherence | Pre-intervention (day 1); during intervention (every 15 days during intervention); after intervention (day 84).
  Adherence level. Adherence will be measured in days of exercise performance by means of a diary questionnaire. Adherence will be coded 0=if on that day they have not done what was prescribed, 1= if they have done some exercise, 2=if on that day they have carried out all the activity prescribed, 3= if they have carried out additional activity.
Engagement | Pre-intervention (day 1); during intervention (every 15 days during intervention); after intervention (day 84).
  Engagement level. Engagement will be measured in days of exercise performance by means of a diary questionnaire. Engagement will be coded 0=if on that day they have not done what was prescribed, 1= if they have done some exercise, 2=if on that day they have carried out all the activity prescribed, 3= if they have carried out additional activity.
Satisfaction level | Pre-intervention (day 1); during intervention (every 15 days during intervention); after intervention (day 84).
  Satisfaction will be measured with a brief interview using a Likert scale. Satisfaction will be recorded on a Likert scale from 0=very dissatisfied to 4=very satisfied.
Incidents | Pre-intervention (day 1); during intervention (every 15 days during intervention); after intervention (day 84).
  Incidents will be measured with a brief interview. The number of incidents and whether or not it has influenced adherence shall be recorded.
Maximum Leg Strength Endurance | Pre-intervention (1 day); after intervention (day 84).
  Maximum leg strength endurance for 30" will be measured with the strength with the 30" Sit-To-Stand (STST). To perform the 30" Sit-To-Stand, from a sitting position, patients will rise and return to the starting position as many times as possible within 30 seconds.
Maximum Arm Strength Endurance | Pre-intervention (1 day); after intervention (day 84).
  Maximum arm strength endurance for 30" will be measured with the 30" Arm Curl Test (ACT). To perform the Arm Curl Test, from a sitting position, as many elbow flexion-extension movements of dominant limb as possible should be performed in 30 seconds with a 2 kg weight.
Submaximum Aerobic Capacity Walking | Pre-intervention (1 day); after intervention (day 84).
  Submaximum aerobic capacity walking for 6 minutes will be measured with the 6-Minutes Walking Test (6MWT). In the 6-Minutes Walking Test, patients are asked to walk the maximum possible distance for 6 minutes.
Post-COVID Functional Status | Pre-intervention (1 day); after intervention (day 84); follow up 1 (3 months after intervention); follow up 2 (6 months after intervention)
  Functional capacity will be measured with the Post-COVID Functional Status Scale (PCFS). In the Post-COVID Functional Status Scale, the levels range from 4 level that means severe functional limitations to 0 that means no limitations and no symptoms."D" level means death.
Depression, Anxiety and Stress | Pre-intervention (1 day); after intervention (day 84); follow up 1 (3 months after intervention); follow up 2 (6 months after intervention).
  Depression, anxiety and stress will be measured with the Depression, Anxiety and Stress Scale (DASS-21). In this scale, each item is answered according to the intensity of each symptom suffered in the last week on a Likert scale from 0 to 3 points. The global scale contains three different blocks for: depression, anxiety and stress. Each block has seven items. The global scale score ranges from 0 to 21 points. In the Depression, Anxiety and Stress Scale, higher scores indicate higher levels of stress, depression and anxiety.
Self-efficacy | Pre-intervention (1 day); after intervention (day 84); follow up 1 (3 months after intervention); follow up 2 (6 months after intervention).
  Self-efficacy will be measured with the General Self-efficacy Scale (GSES).The General Self-efficacy Scale consists of 10 items with a minimum score of 10 points and a maximum of 50 points with Likert-type responses. In the GSES, the higher score indicates higher perceived general self-efficacy.
Behavior in sport | Pre-intervention (1 day); after intervention (day 84); follow up 1 (3 months after intervention); follow up 2 (6 months after intervention).
  Behavior in sport will be measured with the Behavioral Questionnaire in Sport (BRSQ) (36-item version). The Behavioral Questionnaire in Sport measures extrinsic motivation through different factors depending on whether the patient performs physical activity because they believe that it is part of a healthy lifestyle (integrated regulation), because they believe that the activity is important but not pleasant (identified regulation), because of feelings of guilt (introjected regulation) and / or external pressures (external regulation). Intrinsic motivation is measured by three factors, knowledge, execution, and stimulation. Another factor it measures is demotivation. This scale is validated in the Spanish context. Its items are valued using a Likert scale that ranges from 1 (not at all true) to 7 (very true).
Perceived social support | Pre-intervention (1 day); after intervention (day 84); follow up 1 (3 months after intervention); follow up 2 (6 months after intervention).
  Perceived social support will be measured with the Multidimensional Scale of Perceived Social Support (MSPSS). The Multidimensional Scale of Perceived Social Support is validated in the Spanish population by Landeta and Calvete, obtaining high psychometric properties. It is considered a priority scale to be applied in people who are in the process of recovery. It measures social support in three dimensions (family, friends and significant others) and also provides a final score. The version used consists of 12 items that are answered using a Likert scale that ranges from 1 (totally disagree) to 7 (totally agree).
Quality of Life Assessment | pre-intervention (1 day); after intervention (day 84); follow up 1 (3 months after intervention); follow up 2 (6 months after intervention).
  Changes in the quality of life. Quality of life will be measured with the Short Form Health Survey (SF-12-v2). It consists of 12 likert-type items ranging from 1 to 6 points. In the Short Form Health Survey, a higher score indicates a higher self-perceived quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Carolina Jiménez Sánchez, MD, Principal Investigator — Universidad San Jorge; Sandra Calvo, Dr, Principal Investigator — Universidad San Jorge
Locations (2):
- Spain (2):
  - Hospital Real Nuestra Señora de Gracia, Zaragoza
  - Hospital Royo Villanova, Zaragoza

REFERENCES:
- [Derived] Carpallo-Porcar B, Calvo S, Perez-Palomares S, Blazquez-Perez L, Brandin-de la Cruz N, Jimenez-Sanchez C. Perceptions and Experiences of a Multimodal Rehabilitation Program for People With Post-Acute COVID-19: A Qualitative Study. Health Expect. 2025 Jun;28(3):e70283. doi: 10.1111/hex.70283. PMID 40302157
- [Derived] Carpallo-Porcar B, Calvo S, Alamillo-Salas J, Herrero P, Gomez-Barrera M, Jimenez-Sanchez C. An Opportunity for Management of Fatigue, Physical Condition, and Quality of Life Through Asynchronous Telerehabilitation in Patients After Acute Coronavirus Disease 2019: A Randomized Controlled Pilot Study. Arch Phys Med Rehabil. 2024 Aug;105(8):1439-1448. doi: 10.1016/j.apmr.2024.04.014. Epub 2024 May 4. PMID 38710426
- [Derived] Carpallo-Porcar B, Romo-Calvo L, Perez-Palomares S, Jimenez-Sanchez C, Herrero P, Brandin-de la Cruz N, Calvo S. Efficacy of an asynchronous telerehabilitation program in post-COVID-19 patients: A protocol for a pilot randomized controlled trial. PLoS One. 2022 Jul 19;17(7):e0270766. doi: 10.1371/journal.pone.0270766. eCollection 2022. PMID 35853037